# Official study title:

Development of an Adjunctive Video-Based Suicide Prevention Intervention Immediately Following Psychiatric Hospitalization

NCT number: NCT04307394

Document date: 3/28/2022

#### Local IRB # 1910-001 IRBNet #1505531

# BUTLER HOSPITAL INSTITUTIONAL REVIEW BOARD

**PROTOCOL** 

| 1.) Project | |
|---|---|
| Title of Project:Develo | pment of an Adjunctive Video-Based Suicide Prevention Intervention Immediately |
| Following Psychiatric Hospi | talization |
| Principal Investigator (PI): | Lisa Uebelacker, Ph.D. |
| Other Investigator(s): | Brandon Gaudiano, Ph.D., Sarah Arias, Ph.D., Ivan Miller, Ph.D., Lauren Weinstock |
| Ph.D. | |

# 2.) Description of Study

# A. Specific Aims

- 1) Phase 1: We will interview patients (n = 36; Phase 1a) with a history of psychiatric hospitalization for suicidality about their life experiences and coping history. Working with a local film production company, we will invite a subset (n = 12; Phase 1b) of these individuals back to be interviewed on camera for a series of documentary-style videos that will form the basis of *LifePlans*. After the filming of additional clinician-related content, we will create 5, 30-min *LifePlans* episodes using narrative methods. We also will develop an accompanying *LifePlans* workbook using a similar process of feedback and refinement.
- 2) Phase 2: We will conduct an open trial (n=10) to test the feasibility/acceptability of *LifePlans* for hospitalized patients with a pre-admission suicide plan/attempt in the past month. In the hospital, patients will watch the first episode and meet with a hospital social worker, and then watch one episode per week during the first month post-discharge. Patients will be assessed at baseline, and 1- and 6-months post-discharge on suicidal behaviors (primary), suicidal ideation, psychiatric symptoms, functioning, rehospitalization rate, and mechanisms. We will also conduct qualitative interviews with clinical stakeholders (n=12) at mental health hospitals or outpatient treatment centers in the RI area. These clinicians may or may not have treated a patient who participated in the open trial. Stakeholder interview agendas will assess: a) barriers to patients' medication/appointment adherence, b) how the field can use a video intervention to support aftercare, c) challenges patients face upon return to the community post-discharge, d) challenges faced by clinicians/organizations treating individuals with suicidal thoughts and/or behaviors. Modifications will be made to *LifePlans* based on lessons learned from the open trial.
- 3) Phase 3: We will conduct a pilot RCT (n=40) of hospitalized patients (including people enrolled in a partial hospital program) with a recent suicide attempt/plan who will receive treatment as usual (TAU) plus *LifePlans* vs TAU only. We will examine *LifePlans* feasibility and acceptability (video viewing, engagement, satisfaction, recruitment/retention), treatment differences (within relevant confidence intervals) on outcomes (e.g., suicide behaviors), and change on potential mechanisms.

# B. Background

Suicide and attempted suicide are major public health issues in the U.S., accounting for almost 45,000 deaths in 2016, and over 1 million attempts each year. Although recent years have seen significant advances in our

knowledge of efficacious treatments for many psychiatric disorders, the suicide rates in the U.S. have been increasing since 2000. Even with increased efforts in recent years, there still has been a relative paucity of research devoted to developing or testing innovative interventions directly targeting suicidal behavior to reach those most in need. Some treatments (e.g., cognitive behavior therapies) have been found to reduce rates of suicide attempts, but these interventions require substantial training and are lengthy and costly to administer. On the other hand, minimally intensive interventions (e.g., follow-up letters, postcards) have shown mixed results. More efficient and effective "middle ground" interventions developed to prevent suicidal behavior are clearly needed. We urgently need interventions based on evidence-based principles that decrease suicidal behavior and are feasible to deliver to large numbers of patients at times when their risk for suicide is high.

Narrative communication is an alternative strategy for disseminating behavior change principles that has shown efficacy for improving health behaviors. Our own pilot work suggests it may be useful for treating depression. Narrative methods refer to people with lived experience talking about both their struggles and successful ways of coping. Narrative strategies are consistent with social learning theory: people learn by observing others like themselves. An advantage of narrative communication that it is often viewed as more engaging by patients (than didactic communication) and, with the help of video, is easier to disseminate than traditional interventions delivered by clinicians. Narrative communication interventions can be designed to promote key principles from evidence-based psychotherapies.

In this treatment development project, we propose to develop and test a narrative-based video intervention for people with suicidal behavior or plan (with or without intent) being discharged from psychiatric hospitalization. The period immediately following discharge, and the entire year after discharge, is a time of substantially increased risk for suicidal behavior. In response to the need for treatment over this transition, we previously developed a psychosocial intervention, Coping Long Term with Active Suicide Program (CLASP), in which clinicians deliver up to 15 in-person and telephone sessions with patients and families starting during a hospitalization and continuing for 6 months post-discharge. CLASP targets risk factors associated with suicidal behavior (coping strategies, social support, adherence, hopelessness) in order to reduce subsequent risk. Initial research on CLASP is promising, with a 40% reduction in suicide attempts compared to controls over 6 months follow-up.

In this project, we propose to develop a new intervention, called *LifePlans*, based on the CLASP model but using an easily disseminable video-based format in which real patients discuss their history of suicidal behavior and the coping strategies that they used to stay safe. *LifePlans* will consist of 5, 30-min episodes that highlight patients' experiences consistent with the CLASP model. Episodes will cover these topics: 1) developing a personalized "Life Plan" to stay safe and restrict means, 2) clarifying valued life domains and related goals to improve hopefulness, 3) using informal problem solving to cope better with illness, 4) improving communication with family/friends to increase social support, and 5) adhering to primary treatments including pharmacotherapy and psychotherapy to promote illness management. To aid in video content development and planning, we will also conduct qualitative interviews of clinical stakeholders regarding their perspectives on the video series.

#### C. Experimental Method

# **C1. Brief Description of Subjects**

Phase 1: Participants with a history of psychiatric hospitalization for suicide plan and intent or attempt (n=36) will be initially interviewed (Phase 1a), with a subset (n=12) selected to be part of the LifePlans videos (Phase 1b).

Phase 2: Participants currently psychiatrically hospitalized with suicide plan (with or without intent) or recent suicide attempt in the past month (n=10) will receive TAU + LifePlans starting during their hospitalization and continuing after discharge. We also will conduct 30-minute individual interviews of clinical stakeholders (n = 12). Interviews will be led by members of the investigator team and a study research assistant (RA) listening to the conversation and taking notes. Interview agendas will be developed so that

Date most recently revised 3/22/2022

Protocol Version 2.5 

participants will receive similar types of questions, as well as those that may be specific to their job responsibilities (e.g., clinical counselor vs psychiatrist).

Phase 3: Participants currently psychiatrically hospitalized or enrolled in a partial hospital program with suicide plan (with or without intent) or attempt (n=40) will be randomized to receive TAU vs TAU + LifePlans starting during their hospitalization and continuing after discharge.

#### C2. Study Design

# **Phase 1: Development Phase**

The aim of this phase is to develop a brief narrative-based video intervention (LifePlans) for use with hospitalized patients with a suicide intent and plan or suicide attempt prior to admission. Consistent with our own previous work and that of others, 1,2 we will use a research strategy that allows us to elicit compelling participant narratives from a specific community (people with a history of suicide plans/behaviors) that are chosen and framed in order to communicate evidence-based therapeutic strategies. This series of videos will be intended to be adjunctive to treatment from community mental health providers that occurs during the very high risk period of one month post-hospitalization. Ultimately, this type of video program can be one component of a Zero Suicide package as implemented in a health system of care. The five steps to the intervention development strategy are: 1) initial qualitative interviews to identify participants for videorecording (n=36 total); 2) selection of a subset of participants initially interviewed in step 1 for participation in videorecordings; 3) videorecording and editing of the selected participant interviews (n=12 total); 4) stakeholder feedback on video content; 5) professional framing, editing, and workbook creation for final LifePlans intervention. This process will be done in an iterative fashion to allow us to incorporate stakeholder feedback and lessons learned from earlier iterations to finalize the video product and workbook. The first four steps will be repeated three times each in order to yield the final set of videos featuring 12 participant interviews We have previously used this methodology to successfully complete a previous video-based narrative intervention.<sup>3</sup>

# **Development: Recruitment**

We will select participants to interview about their experiences with suicidality and their recovery process. See full inclusion criteria below. Recruitment will occur via advertisements in the community and outpatient mental health settings and in collaboration with community patient support groups. We will also recruit via social media and other online forums. We will attempt to recruit participants who have successfully completed previous CLASP studies who gave us permission to contact them about future studies. Interested participants will be invited to call research staff or will request a call via a secure online format. Staff will describe the goals of the study over the phone and conduct an assessment of inclusion criteria. If they are eligible, we will schedule them for an in-person interview OR a remote video-based interview using a HIPAA compliant online platform, or a phone call if they prefer or don't have access to a computer or smartphone. At the start of that appointment, we will conduct an informed consent process and obtain written OR verbal consent (depending on whether the interview is in-person or remote)

Given our modest goals, we do not anticipate problems with recruitment. However, it is possible that some individuals will not want to be featured in videos that talk about suicide and that will be shown to other people. To address this concern, we will give participants the opportunity to view their completed video (which will portray the participants in a favorable light) and to withdraw the video, or parts of the video, at that time. We will also create the final intervention in such a way that participants may request to withdraw their videos even once they are live, and we will do so. See Human Subjects Phase 1 for details.

#### **Development Step 1. Narrative Collection (Phase 1a)**

We will design an interview guide, and Drs. Gaudiano, Uebelacker, and Arias, and Mr. Audet, will conduct initial 60 min interviews. Based on our previous project, we estimate that we will have to conduct these initial interviews with 36 participants total (12 participants x 3 iterations) to identify 12 (i.e., 4 participants x 3

iterations) who ultimately will be eligible and willing to be videorecorded for LifePlans (in the next step). The interview guide will be designed to elicit experiences of successful coping with suicide-related thoughts, feelings, behaviors, and situations that are consistent with CLASP principles (see next section). For example, we will ask: "Tell me about your experiences coping with suicide thoughts or behaviors." "What have you found works for you?" "Tell me about your experience with psychiatric hospitalization. What was helpful for you when you were leaving the hospital and transitioning home?" We will directly ask about risk factors targeted in CLASP: "What are reasons for living? What important personal values guided your recovery? What kept you going through this crisis?" "What helped you to manage feelings of hopelessness?" "Were there difficult problems you needed to solve when you left the hospital?" "How did friends or family help or not help?" "How has mental health treatment been helpful for you?" "What barriers did you need to cope with to access treatment?" We will audiorecord or videorecord and transcribe interviews. Audio and video will be stored in a secure, CNE-compliant location (See section D2, page 14, for details).

We will also collect self-report information on demographics and current treatment status. Participants will be paid \$40 at this stage.

# <u>Development Step 2. Selection of interviewees for participation in LifePlans video</u>

We will next code interview transcripts based on consistency with the CLASP model. Two members of research team (i.e., the person conducting the interview + one other member of the research team) will code each interview on consistency with the following **CLASP principles** that will be the focus of the video series:

- <u>Hopefulness by clarifying life values and consistent actions</u> (e.g., "I thought about how being a mother was really important to me, and how I could spend more time with my son helping him with his homework);
- Use of <u>problem-solving</u> strategies to cope better with illness including a positive problem-solving orientation (e.g., I wanted to look for a new job, so I first started to update my resume.");
- Improving <u>communication with and support from family/friends</u> and treatment providers (e.g., "When I was feeling like things would never get better, I reached out to my sister and let her know what was wrong.");
- <u>Treatment adherence</u> and engagement (e.g., "In addition to my medication, I decided to give the therapist I was referred to a call to schedule an appointment.");
- Safety planning, use of a safety plan, and discussion of means restriction.

We will also rate interviewees on their overall story-telling ability: Do they tell stories that have a beginning, middle, and end? Are the stories detailed and engaging? Similar to previous work, coders will use a scale of 0 (CLASP-inconsistent); 1 (not present) to 3 (very strong and consistent with CLASP). Discrepancies will be resolved via consensus. Based on these ratings, the study team will choose 12 interviewees total for participation in the LifePlans video. Selection will be based on consistency with CLASP and story-telling ability within the context of ensuring demographic diversity (race, ethnicity, age, gender, sexual orientation) as well as clinical diversity (those with a recent attempt vs. those without) in the ultimate product.

# Development Step 3. Videorecording and editing (Phase 1b)

We will invite the 12 chosen interviewees (4 in each iteration) to participate in a videorecording session. Given that the videos may be widely viewed, one of the PIs or Co-Is will conduct the informed consent process in order to ensure that participants have a full understanding of the process. We will review the American Foundation for Suicide Prevention's (AFSP) "Speaking out about Suicide" guidelines with interviewees before the session (https://www.sprc.org/resources-programs/speaking-out-about-suicide). Next, Mr. Kahn, our expert film producer, will re-interview each of the chosen participants, using the interview guide described above and with input from the investigators about previous statements made by the interviewee that are judged to be important. Interviews will be videorecorded with expert videographers (from FlatIron Works) in order to ensure a high-quality product. Mr. Kahn is very experienced with this approach, and has produced numerous engaging, documentary style videos for hospitals and non-profit organizations. He has previously worked with this research team, and his staff have received human subjects training. He and his staff will complete necessary Butler Hospital paperwork (e.g., HIPAA and independent contractor agreements) to work on the project.

Because some interviewees may not feel comfortable attending an in-person interview, we will also offer an option for remote professional videorecording. After a remote (video or audio) informed consent process, participants will sign all informed consent documents, including acknowledgment that parts of the video produced will be public, on REDCap. The videorecording team will send a package to the participants via mail or deliver it in person that includes a videocamera and other equipment, with instructions for how to set it up. This team has successfully done this process with other people, and can guide participants through the set-up, and then conduct the interview remotely.

Even when the equipment is delivered in person for local participants, the actual interview will still be conducted with the crew outside the participant's home. However, the videographers may need to enter the participant's home briefly to help set up equipment or solve technical issues (e.g., 5-10 minutes) with the participant's permission and with everyone properly masked and socially distanced. The participant will be free to not permit the videographers in the home if they are not comfortable with this.

Next, videographers and investigators will work together to edit video from each person into narrative clips that focus on key CLASP principles (described above) and omit aspects of the interview that are less relevant. We will follow the safe story guidelines set by the AFSP when editing the clips (e.g., avoiding phrases such as "committing suicide" and details about suicide methods). When we have done this previously, this has yielded a series of four to six 3-5 minute "vignettes" for each interviewee. Other video footage is discarded. We will then give participants the opportunity to screen their own video vignettes before moving on to the next step in the research process in order to be sure that participants are comfortable with the dissemination of the video.

#### Development Step 4. Stakeholder feedback

We will screen selected vignettes with the Patient and Family Advisory Council at Butler Hospital in order to get their feedback on the clips. This Council is made up of volunteers who are current or former patients at the hospital, and family members of current or former patients. It meets monthly and provides input on various hospital programs and policies. We will ask members of the Council about engagement in videos or "transportation" (e.g., What aspects of the videos were engaging? What was not engaging or not believable? Do you think that this person has a message that is useful or relevant for patients who are just discharged from the hospital?). We also will ask the Council about video "message": "What did you think was the most important point of the video?" "What might Butler patients learn from this video?". We will audiorecord and transcribe member responses. Lessons learned regarding transportation and message from the Advisory Council may guide: 1) final choice of vignettes to be used in LifePlans; 2) refinement of interview guide for the next iteration; 3) who we choose for future videos; 4) how the videos are further edited; 5) how the videos may be framed and 6) what workbook exercises would be most helpful, understandable, and effective.

# **Development: Repetition of steps 1-4**

We will repeat steps 1-4 three separate times until we have video narratives recorded from 12 individuals. We will divide the video content into 5 separate, 30 min "episodes," with each episode centered on a key CLASP principle: 1) Values Clarification and Goal Setting; 2) Problem-Solving Part 1; 3) Communication with Family, Friends, and Professionals; 4) Problem-Solving Part 2; 5) Communication Part 2. The principles of Treatment Adherence/Engagement and Safety Planning/Means Restriction will be included throughout the five videos. For example, values clarification might naturally lead to means restriction, and one might problem-solve about how to enact means restriction. We will always shoot more video than will actually be used and choose video clips to include based on our conceptual framework. However, if there is other content that that is not directly related to these concepts but seems to be very useful and potentially consistent (even if novel), we will consider including this as supplemental video material.

#### Development Step 5. Professional framing, final editing, and workbook creation

We will write a series of "frames" for the patient narratives consisting of clips in which professionals introduce key concepts, provide background information on patient narratives, and summarize ideas. Professional frames will be written to keep the focus on the patient narratives (rather than on the professional), but highlight key CLASP principles (consistent with the AFSP's safe stories guidelines). We will screen these "professional frames" with the Patient and Family Advisory Council so that we may incorporate their feedback. The patient narratives and professional frames will be combined to develop a series of 5 videos, with each episode being 30 minutes long but divided into smaller sections for ease of viewing and editing.

In addition, we will develop an accompanying workbook or "personal journal" for participants that includes a self-help guide which encourages participants to write about what they learned in the videos and how they will take similar steps in their own lives to cope with suicide ideation/ behavior. In brief, steps will include: 1) eliciting treatment strategies that our initial pool of interviewees report they have found helpful in managing their own suicidality; 2) coding these strategies for consistency with the CLASP model; 3) filming and editing the selected interviewees discussing their use of CLASP-consistent strategies for potential inclusion in the workbook; 4) obtaining stakeholder feedback and refining the strategies to be included in the workbook; and 5) final framing, editing, and creation of workbook content. Through a variety of exercises, they will be encouraged to write their own narrative and life plan. Research demonstrates the potential utility of written emotional disclosure for depression.<sup>4,5</sup>

Exercises include: 1) completing the LifePlan document, 2) guidance on identifying personal values, potential barriers/obstacles, and a plan for engaging in values-consistent actions, 3) guidance on identifying and addressing treatment beliefs/barriers, 4) practice problem-solving to cope with stressors, and 5) developing strategies for effective communication for engaging with friends/family.

# Phase 2: Open Trial

The aim of this phase is to conduct an open pilot study (n=10) to test the feasibility and acceptability of LifePlans in conjunction with treatment as usual (TAU). We will enroll hospitalized patients with a suicide plan/attempt prior to admission in the past month (see full inclusion criteria below). Patients will watch the first episode prior to discharge, and then watch one episode per week during the first month post-discharge. Patients will be assessed at baseline, and 1- and 6-months post-discharge on suicidal attempts and deaths (primary), suicidal ideation, depressive symptoms, functioning, and target mechanisms (i.e., CLASP risk factors). We will examine and seek to improve feasibility and acceptability of LifePlans. Modifications will be made to LifePlans as needed based on lessons learned from the open trial.

# **LifePlans Intervention**

One advantage of video is that it can be made available in multiple formats at low-cost. In order to ensure that watching of the videos is spaced out over time, and to serve as a reminder to watch the videos, we will have the participants watch their first video at baseline (in the hospital) and give them their workbook. This will provide the chance for the interventionist to address any questions they may have about the video. Subsequently, we will send them a link to the first episode at home and encourage them to rewatch it to increase of the "dose" of the intervention. (If a participant prefers, we will send him/her DVDs as an alternative). We will send a one link per week via email to the 2<sup>nd</sup>, 3<sup>rd</sup>, 4<sup>th</sup>, and 5<sup>th</sup> episodes throughout the month after hospitalization. We send the videos separately to spread out the dose of the intervention over the first month as they will be designed to help the patient transition from hospitalization to outpatient care at home. In addition, sending one video per week allows the patient time to fully absorb the message of that video before moving on to the next. Patients will have access to all previous videos; we will encourage them to watch each video twice to improve their understanding.

Between 4-7 days after the patient receives the link to the 2<sup>nd</sup> episode, the study clinician will call the patient to check-in. During the call which will last 10-15 minutes, the clinician will inquire about the participant's perceptions of the videos and encourage them to update their Safety Plan/Life Plan based on what they watched in the videos. If the patient reports suicidal ideation, the clinician will follow the study safety protocol to conduct a risk assessment.

**LifePlans Promotion/Adherence.** Participants will complete brief REDCap surveys after viewing each LifePlans video that will allow us to track adherence. We will send out automated prompts and reminders via

email to increase adherence. At patient discharge, we also will send patients' outpatient clinicians information on LifePlans (along with video links) and update them during the study as to their patients' progress via messages sent using electronic medical records. We will emphasize the importance of use of the workbook during the predischarge session with the hospital interventionist at the start of LifePlans. We plan to develop the workbook in conjunction with our storytelling videos using a similar process involving patient feedback and refinement. We will integrate the workbook exercises into the LifePlans videos to prompt completion.

# Treatment as usual (TAU)

**Butler Hospital.** On the inpatient units, we will include two study interventionists as part of our research team. They will be responsible for checking in with the patient, discussing video content, and answering questions after he/she views the first video as an inpatient. As part of our treatment development aims, these interventionists will provide feedback about integration of video viewing with other therapeutic activities on the inpatient units. Drs. Gaudiano and Uebelacker will meet with the interventionists on a weekly basis.

The average length of stay as a psychiatric inpatient at Butler Hospital is 5-6 days. In the context of the therapeutic milieu, patients receive individual treatment and attend group therapy. Families are included in treatment and treatment planning as appropriate. Additional therapeutic activities include sensory modulation activities, daily exercise, and recreational activities. Patients with suicide risk are involved in a safety planning process prior to discharge. (If a study participant does not have a written safety plan when they enroll in the study, the study interventionist will be responsible for ensuring that this treatment goal is accomplished.)

# **Outpatient Treatment.**

Whenever a patient is enrolled and is receiving LifePlans, we will send the outpatient clinician a note via the EHR or fax describing the patient's participation. The clinician also will be offered links to the videos and workbook, and a summary of each "episode" to inform them about the patient's study participation. This will ensure that the videos serve as an adjunctive treatment, and that patients have the opportunity to discuss videos with a clinician (and vice versa) should they choose to do so. The research team will conduct qualitative interviews with a subset of these clinicians in order to better understand how the videos may be integrated into ongoing outpatient treatment.

# Screening Process and Recruitment (phases 2 and 3)

Our team has developed effective procedures for recruiting from the inpatient milieu (during Phases 2 and 3) as well as the partial hospital milieu (only during Phase 3). We will obtain a Protected Health Information (PHI) waiver for review preparatory to research. Then, we will screen electronic medical records at Butler Hospital to identify potentially eligible participants. Patients meeting inclusion criteria that can be assessed via chart review (i.e., criteria 1, 3, 5), and after obtaining attending physicians' permission, will be approached by research staff. Patients will be approached in-person on the units or if they are attending a partial hospital program virtually, they will be contacted by phone using the number provided in their chart. Staff will provide a description of the study and invite patients to participate in additional screening to determine study eligibility. Those consenting and meeting all inclusion criteria will be invited to participate in the study.

# Research Assessments (phases 2 and 3)

Assessments will be conducted: 1) to assess feasibility and acceptability, uptake, transportation, and understanding of key messages; 2) to assess inclusion criteria; or 3) to pilot outcome measures or potential mediators for the eventual large-scale RCT. See the table below for the purpose of each instrument and the assessment schedule. A trained research assistant will conduct all assessments. After the baseline assessment, we will conduct assessments at 1- and 6-months post-discharge. We will also administer weekly post-video surveys in order to assess completion and acceptability ratings.

**Treatment acceptability/feasibility.** Intervention credibility and patient expectations for intervention success after viewing the first episode will be measured with the <u>Credibility Expectancy Questionnaire (CEQ).</u> 6 The Client Satisfaction Questionnaire (CSQ-8)<sup>7,8</sup> will be used post-treatment to assess satisfaction with interventions. We will also use <u>qualitative</u> responses to a detailed post-treatment interview to gain participants' feedback about interventions and research procedures, including whether there was any contamination

Date most recently revised 3/22/2022 Protocol Version 2.5 between arms, with participants in LifePlans sharing videos or video content with participants in the treatment as usual arm.

We will ask participants to complete additional assessments reflecting the content of LifePlans. Participants will complete video completion surveys of the time that they spend watching the video and the particular sections watched. If they did not watch the videos, participants will answer questions on any barriers that prevented them from watching. To assess transportation/engagement, we use a modified version of the Transportation Scale 9 (11 items) we previously developed that is appropriate for watching a video. Sample items include: "The [video about XX] affected me emotionally" or "I found my mind wandering while [watching the video about XX.]" Items are rated from 1 "not at all" to 7 "very much." The total scale score is calculated by taking the average of all items. In addition, participants will complete a Video Acceptability Scale, which is adapted from a 7-item Likert-scale measure (1=not at all and 7=very much) designed for technology-assisted interventions by Ondersma et al. 10 that assesses how participants feel about their experience: overall liking, interesting, ease of use, understandable, respectful, or annoying. To assess message understanding, we will use a Message Scale, which consists of questions designed to: 1) enhance the impact of the intervention; and 2) provide data to us about their reactions to the video. The questionnaire includes these questions: 1) What did you like about this video? What did you not like about this video?; 2) What was the main message that you got from watching this video?; 3) Does this video have any relevance to your life? What relevance does it have to your life?; and 4) What might you do differently as a result of watching this video? We will use qualitative data analysis techniques to analyze participants' responses.

| | Purpose | Timepoints |
|---|---|---|
| Freatment Acceptability, Feasibility, Uptake, Transportation | | <u> </u> |
| Credibility Expectancy Questionnaire | Р | BL |
| Client Satisfaction Questionnaire | P,O | M1 |
| Qualitative Interview | P | M1 |
| Video Completion Surveys | P | W1, W2, W3, W4 |
| Fransportation Scale | P | M1* |
| Video Acceptability Scale | P | M1* |
| Message Scale | P | M1* |
| Psychiatric Symptoms and Functioning | | |
| Columbia Suicide Severity Rating Scale | 0** | BL, M1, M6 |
| Modified Scale for Suicide Ideation- | 0 | BL, M1, M6 |
| PROMIS-29 | 0 | BL, M1, M6 |
| PROMIS Depression Short Form*** | 0 | W1, W2, W3, W4 |
| Hospital chart review | I,O | BL, M6 |
| Psychosis Screening Questionnaire | 1 | BL |
| Mental Help Seeking Attitudes Scale | 0 | BL, M1, M6 |
| Personal Suicide Stigma Questionnaire (self-blame subscale only) | 0 | BL, M1, M6 |
| Potential Mechanisms (CLASP Targets) | | |
| Multidimensional Scale of Perceived Social Support | Med | BL, M1, M6 |
| Brief COPE | Med | BL, M1, M6 |
| Valuing Questionnaire | Med | BL, M1, M6 |
| Treatment Utilization | | |
| Freatment History Interview | | BL, M1, M6 |
| Outpatient and Hospital Chart Review | | BL, M1, M6 |

**Note.** Purpose: P=Pilot study target outcome; O=Outcome in large-scale RCT; I=Inclusion criteria; O\*\*=Primary outcome in large-scale RCT; C=Characterize sample; Med=Potential mediator in a larger scale RCT. Timepoints: BL=baseline; W1, W2, W3, W4=Week 1, 2, 3, and 4 of the intervention. M1 and M6=Month 1 and 6. M1\*=M1 during the pilot RCT, but weekly during the open trial.\*\*\* The PROMIS Depression Short Form was added for the pilot RCT.

**Suicidal Behaviors.** The Columbia Suicide Severity Rating Scale (C-SSRS) <sup>11</sup> will be used to assess suicide ideation, intent, plans, and behavior. C-SSRS interviews will be conducted by trained research staff supervised by Dr. Uebelacker with consultation from Drs. Miller and Weinstock. Training procedures consist of: a) review of written materials, b) didactic instruction; c) practice interviews with review and feedback from senior staff; and 4) continued practice, training and feedback until high agreement with established consensus ratings are met (e.g. 3 consecutive C-SSRS ratings are within 2 points of our consensus ratings). We will assess interviewers'

reliability in an ongoing manner. Following initial training, interviewers and senior staff meet on a monthly basis to review tapes, address questions/issues, and monitor interrater reliability.

To ensure that we capture as much suicide-related data as possible, we will utilize procedures that have been developed for current ongoing large-scale suicide prevention clinical trials led by Dr. Miller (RO1 MH101129) and Dr. Weinstock (U01 MH106660). We obtain releases of information from patients at study start to conduct chart reviews throughout the study covering the two major healthcare systems in RI (CNE and Lifespan) and their corresponding EDs and inpatient units. We also collect treatment utilization data via self-report (THI) during follow-up assessments, and, at that point, we can ask participants for releases of information to request discharge summaries from additional hospitals that the patient may report attending. Consistent with previous studies, we scrutinize all hospitalizations or ED visits with any of the following characteristics: evidence of self-injury, mental health concerns, ingestion/overdose, and traumatic injury. Staff then read the discharge summary to determine if there is any evidence of current or recent intentional self-harm ideation or behavior, including whether any injury is sustained. Staff also use carefully developed definitions of suicide ideation and suicide attempt (from C-SSRS criteria) to determine whether there is evidence of either event in the medical record.

If the patient dies, staff record the death and whether there was any evidence of intentional self-injury leading to the death. As we have done in previous studies, if we are unable to locate a participant at follow-up, we will state or national death registries to ascertain whether he/ she died, and if so, cause of death. Thus, suicide outcomes will be determined using all data collected during the study from all possible sources, including follow-up assessments (C-SSRS), b) hospital chart reviews, c) and community clinician reports. Data from all sources will be reviewed by two research team members for congruence. Note that we will obtain releases of information from patients at study start to conduct chart reviews throughout the study covering the two major healthcare systems in RI (CNE and Lifespan) and their corresponding EDs and inpatient units. Disagreements between raters will be reviewed and adjudicated by Drs. Gaudiano (MPI) and Arias (Co-I). All reports will be classified using C-SSRS criteria. In a larger-scale clinical trial, our primary outcome will be a composite: a) suicide attempts or b) suicides.

Other Symptoms. We will use the following self-report scales: the Modified Scale for Suicide Ideation (MSSI)<sup>13</sup> which provides a score indicating overall severity of suicide ideation; and the PROMIS-29, which assesses pain intensity on seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance). We will also have participants in both study conditions complete the PROMIS Depression Short Form each week of the intervention to assess depressive symptoms. In addition, we also will assess the change in distress and perceived helpfulness during each week of the intervention for those assigned to LifePlans: 1) how distressed participants felt while watching the videos (5 point scale from "more distressed" to "less distressed"), 2) how distressed they felt after watching the videos (5 point scale from "more distressed" to "less distressed"), and 3) how helpful they felt the videos were (5 point scale from "very unhelpful" to "very helpful"). In order to ascertain inclusion criteria, we will use chart review and the Psychosis Screening Questionnaire<sup>31</sup> to screen out people at baseline. Finally, we will use the self-blame subscale on the Personal Suicide Stigma Questionnaire (PSSQ) which is a self-report measure that has been found to be reliable and valid for assessing stigma in persons who have suicidal behaviors.

**Potential Mediators.** Potential mechanisms will be assessed using the following self-report scales: the Multidimensional Scale of Perceived Social Support (MSPSS)<sup>21</sup>, which is a reliable and valid measure of 3 aspects of social support (family, friends, and significant other); the <u>Brief Cope</u><sup>22</sup>, which assesses strategies used for coping in response to negative life experiences; and the <u>Valuing Questionnaire</u> (VQ) which is a reliable and valid measure that assesses the extent to which a person lives by their values.

**Potential Moderators**. We have identified several potential moderators of CLASP effects in our previous research that we believe may also be relevant to the proposed project, which we will consider testing in future, larger-scale studies. The manuscript describing these results is currently in preparation. The following factors were found to moderate the effects of CLASP in the previous ED-SAFE study (U01 MH088278) and are also potentially relevant to LifePlans: marital status (CLASP more effective for those not married) and number of previous psychiatric hospitalizations (CLASP more effective for those with more hospitalizations). We will also consider whether recent suicide attempt status and lifetime suicide attempt status moderates outcome.

**Treatment utilization.** We have adapted a brief, structured Treatment History Interview (THI)<sup>25</sup> which allows

us to collect information about other depression treatments such as inpatient hospitalization or psychotherapy, including any care that happens outside of the CNE system. We will combine this with information from the outpatient chart review (i.e., from the Providence Center) and inpatient chart review (from Butler Hospital) to gain a full picture of treatment utilization.

Clinical stakeholder interviews. Basic demographic information will be collected from all participants using a short self-report measure. These data will include age, gender, ethno-racial background, education level, duration of employment in current position, and duration of employment in the field. Participants will complete a 30-minute individual interview by telephone or videoconference. Prior to the interview, we will send participants a brief description of the video series and sample content. This interview will be scheduled at the participant's convenience and will be audio or video recorded. Stakeholder interview agendas will assess: : a) barriers to patients' medication/appointment adherence, b) how the field can use a video intervention to support aftercare, c) challenges patients face upon return to the community post-discharge, d) challenges faced by clinicians/organizations treating individuals with suicidal thoughts and/or behaviors. Questions will be delivered in an open-ended format to allow participants to share their opinions.

#### **Retention and Adherence**

We will use several strategies to increase retention for assessments. Research staff will remind participants about appointments, maintain a list of locator contacts for each participant, reach out to contacts as needed, schedule assessments regardless of intervention participation, and have flexibility in when assessments are scheduled. Finally, we will provide transportation if needed for appointments.

# Phase 3: Pilot RCT

The aim is to conduct a pilot RCT (n=40), with participants randomized to treatment as usual (TAU) or TAU + LifePlans. We will enroll hospitalized patients with a suicide plan/attempt prior to admission in the past month (see full inclusion criteria below). Methods will be similar to those described in the open trial (see previous section for Phase 2), with only the differences noted below. We will continue to focus on acceptability and feasibility, including an evaluation of the proposed research design.

#### Phase 3: Control condition description and rationale

The control condition will be TAU, which, as noted above, will include Hospital Safety and Discharge Planning as part of inpatient care, followed by outpatient care at a CNE outpatient site. In choosing TAU as a control condition, we considered the nature of the LifePlans intervention. LifePlans is designed to be adjunctive to TAU and in fact to encourage adherence to outpatient treatment plans developed in the hospital. We did not choose a more robust control condition because LifePlans is designed to be a lower-intensity intervention (thus increasing its potential reach) and not to replace existing treatments (but, in fact, to enhance them).

#### **Phase 3: Randomization**

Participants will be randomized using a 1:1 ratio to either TAU or TAU + LifePlans. Randomization will be stratified by: a) gender (male/ female/ non-binary) and b) suicide attempt vs. plan prior to admission. Treatment arm assignments will be blocked in blocks of 4 or 6 participants (randomly ordered). A staff member with no other study responsibilities will set up randomization tables in REDCap, and other research staff will not have access to the tables. Participants will be randomized following the baseline assessment using the randomize feature in REDCap. This ensures allocation concealment.

#### **C3. Specific Procedures or Treatments**

See C2. Study Design.

# C4. Data Analysis

This pilot study has the primary aims of refining interventions and research procedures for a subsequent RCT to test the efficacy of LifePlans. In the past, researchers have used pilot data to estimate an effect size to assist in future power calculations. Kraemer et al.<sup>26,27</sup> emphasized the limitations of this practice due to the likelihood of large standard errors surrounding effect size estimates, and the concern that RCTs should be powered to detect a difference between groups that is considered to be a minimally clinically significant difference. In light of these concerns, we propose the following analysis plan.

# **Target treatment development outcomes**

We will use descriptive statistics to summarize all variables. At the end of the open trial, and midway and at the end of the pilot RCT, we will examine acceptability and satisfaction outcomes for LifePlans and for the overall study. When the outcome is not met, the research team will investigate and discuss the issue, and depending on the perceived reasons for the discrepancy, may modify relevant research procedures to address the issue. For example, if uptake is low, we will try to modify instructions to participants in order to increase uptake.

#### Qualitative data analyses

This is a mixed methods study and requires the use of qualitative data analytic techniques to understand feedback from qualitative interviews in the open trial and pilot RCT (section C3.6), and to code the Message Scale. For post-treatment interviews, and clinician interviews, we will audiorecord and transcribe interviews, and use a template organizing style to analyze these data.<sup>28</sup> That is, using an iterative approach, Dr. Uebelacker will develop a codebook with categories of responses. After the team codes 3-5 interviews together, and further refines the codebook, all members of the investigative team will separately categorize quotes from the additional transcripts using qualitative data analysis software (atlas.ti). Then the entire research team will meet to review quotes and categories, and differences of opinion will be resolved via consensus. If necessary, new categories will be developed.

For the Message Scale, we will train two research assistants who are otherwise unconnected with this study to use a coding system. They will independently code all responses; 25% of responses will be coded by both research assistants in order to examine inter-rater reliability. For each of the key CLASP principles, coders will use a scale of 0 (CLASP-inconsistent); 1 (not present) to 3 (very strong/ consistent) to code responses on the key CLASP elements. To be considered to have understood the intended message, participants must have a score of "2" or greater on at least 2 of the key CLASP elements.

# Change over time

In the open trial, we will examine within-group changes over time (from baseline to 1-month and baseline to 6-month), on suicide outcomes including attempts and deaths, psychiatric symptoms, psychosocial functioning, rehospitalizations due to suicide behavior, and potential mechanisms. In the pilot RCT, we will also use effect size estimates to characterize group differences on these outcomes at 1- and 6-month follow-ups. We will calculate 95% confidence intervals (CIs). Because the CIs will likely be large, these analyses may not permit definitive conclusions. Given the limitations and goals of small n studies, we hope to build our case for a future full-scale RCT by focusing primarily on the feasibility, acceptability of LifePlans and of the research design. Some parameters estimated in this pilot study (e.g., stability of outcome measures across timepoints) will be used to generate empirical power estimates for a large scale, adequately powered RCT.

## **Power**

Our primary aim in the current study is to examine treatment development variables (acceptability, feasibility, uptake, message) to inform a future full scale trial, rather than to power the study for certain p values. In future studies, we will base power on a minimally clinically significant effect size. For example, in our previous study of CLASP vs. TAU for people transitioning from inpatient to outpatient treatment, we found that, during the 6 month follow-up period, subjects assigned to CLASP in our pilot studies had lower rates of suicide attempts compared with TAU: 8.3% vs 21%, OR=2.77 (95% CI=0.71-10.76). In the context of suicide prevention, these effects are within the range reported for other efficacious interventions. Although LifePlans

Date most recently revised 3/22/2022 Protocol Version 2.5 has a different format, it is based on similar principles as CLASP.

# D. Material Inducements

**Phase 1:** Participants completing the interview phase (n = 36) will receive \$40, mailed to them by check, or (when available) gift card. The subset (n = 12) of participants who complete the video recording will be compensated \$75.

**Phase 2:** For the open trial (n = 10), we will pay participants for assessment interviews: \$20 for baseline, and \$40 for Month 1 and 6 assessments (up to \$100 total). We will also provide transportation if needed for appointments. For the clinician stakeholder interviews (n=12), we will pay participants \$50 for completion of the interviews.

Phase 3: Similar to Phase 2, for the pilot RCT (n = 40), we will pay participants for assessment interviews: \$20 for baseline, and \$40 for Month 1 and 6 assessments (up to \$100). We will also pay participants \$5 for each weekly survey they complete (up to \$20 total). Therefore, they may receive up to \$120 total for their participation. We will also provide transportation if needed for appointments.

#### E. Training of Research Personnel

All study staff will have undergone mandatory online education in human research participants' protection. Pls and research assistants will have training in Good Clinical Practice via an online program. All study staff will undergo specific training relevant to their study roles and responsibilities. Training will be documented via collection of training certificates.

## 3) Human Subjects

#### A. Subject Population

Phase 1: Participants (n=36) will be initially interviewed, with a subset (n=12) selected to be part of LifePlans videos. Participants must meet the following criteria:

- 1. Have a history of psychiatric hospitalization for suicide plan and intent, or attempt;
- 2. Be aged 18 or older;
- 3. Agree that they have developed strategies for successful coping with suicide-related thoughts, feelings, behaviors, and situations;
- 4. Deny current active suicidal ideation or recent (past 3 month) behavior.
- 5. No current significant substance use (defined by Alcohol Use Disorders Identification Test (AUDIT) score <8 <sup>29</sup>; Drug Use Disorders Identification Test (DUDIT)<sup>30</sup> score <8 if only substance used is marijuana; DUDIT score < 6 for males and < 2 for females for any other substance)
- 6. No current psychotic symptoms (defined by a positive answer to any item on the Psychosis Screening Questionnaire <sup>31</sup>)

Phase 2: Participants (n=10) will receive TAU + LifePlans starting during their hospitalization and continuing after discharge.

- 1. Current psychiatric hospitalization with recent (past month) suicide plan (with or without intent), or a suicide attempt within 48 hours prior to hospitalization, as indicated on the hospital chart and confirmed by administration of the C-SSRS <sup>11</sup>. Specifically, on the C-SSRS, this is operationalized to a "yes" on item 3, 4, OR 5, AND/OR a "yes" to suicide attempt/ interrupted attempt/ or aborted attempt.
- 2. Ability to speak, read, and understand English well enough to complete the procedures of the study.
- 3. Aged 18 or older.
- 4. Regular access to a means of watching videos, i.e., a smartphone, tablet, computer, or DVD player.

Date most recently revised 3/22/2022 Protocol Version 2.5

- 5. No current psychotic symptoms (based on chart review and the Psychosis Screening Questionnaire)
- 6. Plan to continue outpatient treatment.

We also will select clinical stakeholders (n=12) for participation. Inclusion criteria are: (1) age 18 or older, and (2) works as a clinician in a mental health program or facility providing services to patients with suicidal thoughts and/or behaviors.

Phase 3: Participants (n=40) will be randomized to receive TAU vs TAU + LifePlans starting during their hospitalization and continuing after discharge.

Participants must meet the following criteria (same as Phase 2):

- 1. Current psychiatric hospitalization with recent (past month) suicide plan (with or without intent), or a suicide attempt within 48 hours prior to hospitalization, as indicated on the hospital chart and confirmed by administration of the C-SSRS <sup>11</sup>. Specifically, on the C-SSRS, this is operationalized to a "yes" on item 3, 4, OR 5, AND/OR a "yes" to suicide attempt/ interrupted attempt/ or aborted attempt.
- 2. Ability to speak, read, and understand English well enough to complete the procedures of the study.
- 3. Aged 18 or older.
- 4. Regular access to a means of watching videos (i.e., a smartphone, tablet, computer, or DVD player) in the place they expect to live after discharge.
- 5. No current psychotic symptoms (based on chart review and the Psychosis Screening Questionnaire)
- 6. *Plan to continue outpatient treatment.*

No minors, prisoners, fetuses/neonates, or decisionally/ cognitively impaired individuals will be recruited.

#### **B.** Recruitment and Consent Procedures

Phase 1a: Recruitment will occur via advertisements in the community and outpatient mental health settings and in collaboration with community patient support groups. We will also recruit on social media and other online platforms. We will attempt to recruit participants who have successfully completed previous CLASP studies who gave us permission to contact them about future studies. Interested participants will be invited to call research staff or will request a call via a secure online format. Staff will describe the goals of the study over the phone and conduct an assessment of inclusion criteria. If they are eligible, we will schedule them for either a) an in-person interview or b) a remote video-based interview using a HIPAA compliant online platform, or c) a phone call if they prefer or don't have access to a computer or smartphone.

If we scheduled an in-person interview, we will obtain written informed consent at that interview.

If we schedule a **remote video-based interview**, with the participant's verbal permission (see attached script; answers to questions in script will be recorded in REDCap), we will email them a link to our video meeting as well as a REDCap link that will bring them to a copy of the Phase 1a consent form that they will be able to use to follow along as we conduct the consent process with them at the beginning of that video meeting. If we schedule a **phone call**, we will send them a copy of the Phase 1a consent form via mail.

At the start of the next appointment (i.e., the video meeting on the HIPAA compliant online platform or the phone call), we will conduct an informed consent process for this study, reviewing the consent document that we sent the participant. We will audio/video record their verbal consent as described in the consent document.

Once we have obtained informed consent, we will start the assessment interview. With participant's permission, we will audio- or videorecord this interview. Audio and video recordings will be stored in a secure, CNE approved location (See section D2, page 14, for details).

Phase 1b: We will invite a subset of 12 chosen interviewees to participate in a subsequent videorecording session with professional videographers. At that point, we will re-consent these participants, and ask them to

sign, in addition to the study consent form, a) a Media Release; b) Public Disclosure; and c) COVID acknowledgement (for as long as COVID remains a risk). We will send these forms to participants ahead of time, and a research staff member will offer to schedule a phone call to go over each form in depth, by phone, so as to minimize time in-person. Participants will then be asked to sign consent and release forms once they arrive for their in-person visit. At that point, given that the videos may be widely viewed, one of the PIs or Co-Is will briefly review the consent documents and answer any remaining questions to ensure that participants have a full understanding of the process.

We will also offer the option for remote professional videorecording. This will follow similar steps to the inperson video recording, and will include:

- 1. Participants will be sent REDCap links to consent documents
- 2. A study PI or co-I will have an audio or video call to review the study and consent documents, including the study consent form, Media Release, and Public Disclosure.
- 3. Videographers will mail a package to the participant that includes a camera and other items needed to set up the videography session.
- 4. Videographers will help the participants with set-up in their homes, and then conduct the session. A study staff member will also observe remotely.
- 5. Participants will then mail the equipment back to the videographers.

Phases 2 and 3: With a HIPAA waiver (see below) we will screen medical records at Butler Hospital to identify potentially eligible participants. Patients meeting inclusion criteria that can be assessed via chart review (i.e., criteria 1, 3, 5), and whose attending physician does not mark as ineligible for research, will be approached by research staff. Patients will be approached in-person on the units or if they are attending a partial hospital program virtually, they will be contacted by phone using the number provided in their chart. Staff will provide a description of the study and invite patients to participate in screening to determine study eligibility. Those consenting and meeting all inclusion criteria will be invited to participate in the study.

For the clinical stakeholder interview during Phase 2, we will consult with our investigator team to identify appropriate clinical stakeholders to approach about study participation. Once identified, Drs. Gaudiano or Uebelacker or another member of the research team will contact the stakeholder directly to introduce the study. If interested, the participant will be mailed or emailed (via REDCap link) a copy of the Stakeholders Informed Consent form in addition to a brief description of the video series. The participant will then be consented over the phone or via videoconferencing. The consent process will be documented either through audio or video recording or via electronic REDCap signature.

For Phase 3, some patients attend the partial hospital programs remotely and cannot be consented in person. With the participant's verbal permission (see attached "Verbal Consent (by Phone) for Use of Email and Videoconferencing"; answers to questions in script will be recorded in REDCap), we will send them a link for videoconferencing (i.e., video meeting on the HIPAA compliant online platform). In addition we will send a REDCap link that will bring them to a copy of the Phase 3 consent form that they will be able to use to follow along as we conduct the consent process with them at the beginning of that meeting. If we schedule a phone call, we will send them a copy of the Phase 3 consent form via email REDCap link. At the start of the meeting, we will conduct an informed consent process for this study, reviewing the consent document that we sent the participant. Participants will answer the questions and electronically sign the consent form in REDCap.

# C. Potential Risks

Potential risks include coercion, discomfort or increased distress due to study procedures, suicide ideation or behavior, and breach of confidentiality. See information below about risk level and impact to subjects.

# D. Protection of the Subject

# **D1. Measures to Minimize Potential Risks**

#### Coercion

<u>Description.</u> Participants could feel that they must participate in the study or, once enrolled, continue to participate.

Risk Level and Likelihood. This is a serious risk but the likelihood of it occurring is judged to be minimal.

Minimization. The risk of coercion will be minimized by following standard procedures for obtaining informed consent. We will fully explain the study procedures, risks, benefits, and alternatives to all patients. Also, patients who do not consent or who withdraw at any time will receive usual clinical treatment with no prejudice. Participant remuneration will be set at modest monetary levels as used in similar studies. In Phases 2 and 3, we will obtain permission form the patient's treating physician to ensure that approaching the patient for research participation is clinically appropriate.

#### Discomfort or increased distress due to study participation

<u>Description.</u> Some participants may find that they feel discomfort or distress in response to completing study assessments or interviews, or when watching LifePlans videos.

<u>Risk Level and Likelihood.</u> This may occur for some participants. Based on our previous experience with this population, we believe that any distress that occurs is likely to be minor and transient.

Minimization. During assessments, research staff will remind participants that they may refuse to answer any question or take a break at any time. Participants will also be reminded that they can choose not to watch a video if they find it too distressing. We will encourage participants to inform research staff if a study procedure is distressing. Finally, we will also encourage participants to talk with their outpatient mental health providers if they find that they are experiencing increased distress for any reason. We will provide referrals to outpatient providers if any participants would like them.

#### Suicide ideation or behavior or psychiatric hospitalization

<u>Description.</u> Participants may reveal active suicide ideation/ plan/ intent/ or behavior during the course of a research interview.

<u>Risk Level and Likelihood.</u> These events may occur in a portion of enrolled participants, particularly in Phases 2 and 3. However, it is very unlikely that these events will be related to study participation.

Minimization. Suicide ideation and behavior, and psychiatric hospitalization, will be monitored via assessment interviews and chart reviews. In assessments, study staff will inquire about suicidal ideation and behavior using the C-SSRS. If any patient reports suicidal ideation, plans, or behavior during the study assessments or other study contacts, the action we will take is dependent on whether the participant is inpatient or he/ she is being treated as an outpatient. If the patient is inpatient, research staff will notify the treating clinician on the inpatient unit, so he/she is aware of the risk reported by the patient. If the patient is outpatient, at the time that suicidality and/or clinical deterioration is identified, a study clinician will immediately evaluate the participant. In such cases, research staff will immediately contact one of the Principal Investigators, Drs. Uebelacker or Gaudiano, or one of the Co-Is, Drs. Miller or Weinstock. All are

licensed clinical psychologists; one of the MPIs or Co-Is will be on call at all times. The clinician will conduct a suicide risk assessment. Depending upon the specific situation, steps taken to ensure a participant's safety may involve: (1) escorting the patient to the hospital's ER for evaluation by an independent clinician and possible hospitalization, (2) alerting inpatient staff to the patient's level of risk, (3) notifying the patient's outpatient clinician(s) at CNE for whom we have releases of information, or (4) calling the appropriate police departments. We will follow the protocol outlined in the DSMP for reporting SAEs to the IRB and other monitoring entities.

# **D2. Measures to Ensure Confidentiality**

<u>Throughout this protocol, we use the term "secure, CNE-compliant location" for storage of electronic files.</u> This refers to the following options:

- CNE research server
- CNE instance of REDCap
- CNE instance of HIPAA-compliant Box
- CNE computer (i.e, password-protected)
- Password-protected, encrypted (128 AES bit or higher) storage device (e.g., audiorecorder, hard drive)

Potential risks due to loss of confidentiality will be minimized by having all information collected and handled by research staff from this study trained to deal appropriately with sensitive clinical issues. All information will be treated as confidential material and will be available only to research and clinical staff. All data collected will be kept in a CNE-compliant location. Patient identifying information will be stored in a separate database and will be password protected. Any paper files with any identifying information will be kept in a locked filing cabinet. No subject will be identified in any report of the project.

In Phase 1b, which includes work with professional videographers, at the earliest possible time after capturing video and/or audio content concerning a research subject or subjects, we will move the content from the camera's memory, storage, SD Cards, etc. to a <u>secure, CNE-compliant location</u>. Once moved, the content will be immediately deleted from the camera's memory, storage etc. This should usually occur within 48 hours of obtaining the content. Audiorecorders and videocameras will be kept in a locked location (e.g., drawer, filing cabinet) except when being used or transported.

Audio/video recordings will be stored on a secure, CNE-compliant location as defined above. Video recordings collected by videographers (consultants) in Phase 1b will be stored on a secure external storage device that is encrypted and password protected per CNE standards (128 bit AES encryption or higher). Once the videographers have completed their work, this storage device will be given to the study investigators. External consultants (videographers) will receive education in Human Subjects (e.g., CITI training) and will also sign a Business Associates Agreement. At the conclusion of the project, any video footage not used in the final product will be destroyed.

Participants in Phase 1 who are chosen to be filmed to be part of the LifePlans videos will be re-consented immediately prior to the time when the raw footage will be shot. Participants will be informed that once the final product is completed and made available to study participants or patients via a web-hosting site on the internet, CNE will no longer have complete control over the video. After the raw footage is shot and edited, participants will have an opportunity to view any footage of them that may be used in the final LifePlans video. At that point, they may request that part or all of the footage not be used in the LifePlans videos, and we will respect their wishes and not use that footage. If participants wish for their videos to be withdrawn at a later date, i.e., after they are hosted on a website, we will make every effort to withdraw those videos from the website. However, in the consent process, we will make it clear that we cannot guarantee that the video has

not been copied by an external party, as the copying could occur even though we will take available measures to prevent it.

## D3. Data Safety Monitoring Plan

## A. Data safety and storage.

Please see section D.2 above.

#### B. Data access.

Only study staff will have access to data. No confidential information may be released outside Butler Hospital without the express written consent of the study participants, unless mandatory for child and elder abuse and in situations in which the risk of suicide or homicide is imminent.

#### C. Educational training.

Please see section on training of research personnel above.

# D. Adverse events and unexpected problems.

The MPIs and Co-Investigator Dr. Arias will be responsible for monitoring and reporting adverse events. They will meet with staff weekly to review any adverse events.

#### **Definitions**

**Serious Adverse Events.** An adverse event (AE) is any untoward medical occurrence in a subject during participation in the clinical study or with use of the experimental agent being studied. A serious adverse event (SAE) is one that meets one or more of the following criteria:

- Results in death
- Is life-threatening (places the subject at immediate risk of death from the event as it occurred; includes a suicide attempt or drug overdose)
- Results in inpatient hospitalization or prolongation of existing hospitalization
- Results in a persistent or significant disability or incapacity
- Results in a congenital anomaly or birth defect

An important medical event that may not result in death, be life threatening, or require hospitalization may be considered an SAE when, based upon appropriate medical judgment, the event may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.

# In this study, we will monitor and report on the following SAEs:

- Suicide behavior
- Inpatient hospitalizations that are:
  - o Suicide-related or
  - Psychiatric in nature or
  - Due to substance use or overdose

Date most recently revised 3/22/2022

Protocol Version 2.5 

• Death for any cause

**Unanticipated Problems (UPs).** The Office for Human Research Protections (OHRP) considers unanticipated problems involving risks to subjects or others to include, in general, any incident, experience, or outcome that meets **all** of the following criteria:

- Unexpected in terms of nature, severity, or frequency given (a) the research procedures that are
  described in the protocol-related documents, such as the IRB-approved research protocol and
  informed consent document; and (b) the characteristics of the subject population being studied;
- Related or possibly related to participation in the research ("possibly related" means there is a
  reasonable possibility that the incident, experience, or outcome may have been caused by the
  procedures involved in the research); and
- Suggests that the research places subjects or others at a greater risk of harm (including physical, psychological, economic, or social harm) than was previously known or recognized.

# **SAE Monitoring and Reporting**

Given that we are recruiting a hospitalized sample with suicide risk and possible substance use disorders, we expect serious adverse events to occur, including suicide attempts, non-suicidal drug overdoses, and psychiatric rehospitalizations,. However, given the nature of the study, it is unlikely that SAEs will be related to the study procedures. If any of these adverse events occur, or any other unanticipated problems are identified, the following procedure will be activated: the research staff member who observes or is notified of an adverse event (e.g., suicide attempt) will notify the MPIs or their designee immediately. All study staff will be educated on the definition of SAEs and UPs so that they may report them to the MPIs as soon as possible after becoming aware of the occurrence of an SAE or UP. We will systematically assess for adverse events throughout the course of the trial (for Phase 2 and 3) via patient interview (C-SSRS, THI) and chart review at Baseline, Month 1, and Month 6. In addition, if a patient reports one of the above SAEs at any time, we will record and review it. The MPIs or their designee will complete an Adverse Event Form for each event that will include a level of severity and determine attribution (intervention-related or not). Reporting timeframes will vary by SAE type. Please see the table below for more details.

| Data type | Frequency of review | Reviewer |
|---|---|---|
| SAEs (expected OR unrelated, including psychiatric | Per occurrence | MPIs (within 72 hours) |
| rehospitalizations and suicide | | Reported to SMC in bi-annual |
| attempts) | | reports |
| | | Reported to NIH in annual |
| | | progress reports |
| SAEs (related) | Per occurrence | MPIs (within 72 hours) |
| | | Reported to IRB and SMC within |
| | | 10 days |
| | | Reported to NIH in annual |
| | | progress reports |

| All deaths | Per Occurrence | MPIs (within 72 hours) Reported to IRB, SMC, NIH within 5 days |
|---|---|---|
| UPs | Per Occurrence | MPIs (within 72 hours) |
| | | Reported to IRB and SMC within |
| | | 10 days |
| | | Reported to NIH in annual |
| | | progress reports |

# **Interim Analysis and Stopping Rules**

There is no interim analysis planned.

This study will be stopped prior to its completion if: (1) the intervention is associated with adverse effects that call into question the safety of the intervention; (2) difficulty in study recruitment or retention will significantly impact the ability to evaluate the study endpoints; (3) any new information becomes available during the trial that necessitates stopping the trial; or (4) other situations occur that might warrant stopping the trial.

#### **Safety Monitoring Committee**

We will appoint a Safety Monitoring Committee (SMC) for trial monitoring. This will be composed of three independent experts with relevant experience. They will receive reports and convene meetings for this study on a twice-yearly basis. They will also receive reports per occurrence of SAEs as described in the table above.

#### **E. Potential Benefits**

**Phase 1:** Benefits to the participant may include satisfaction with having a chance to tell one's story, talk about successful coping strategies, and potentially help other people.

Phases 2 and 3: For all participants in Phases 2 and 3, we will conduct research assessments 1-month and 6-months post-hospitalization. If we identify risk for suicide at those assessments, we will work with participants to ensure that they receive appropriate treatment. Benefits to the participants receiving the LifePlans intervention may include education about and increased motivation for use of coping skills in the following areas: identification of life values and implementing values-consistent behavior; problem-solving strategies; communication with family, friends, and treatment providers; treatment adherence and engagement; and safety planning and means restriction.

All phases/ knowledge to be gained: This study will allow us to develop and pilot test a video-based self-help intervention for use at the high-risk time period of transition from psychiatric hospitalization to community outpatient treatment. We will assess acceptability, feasibility, and safety of this intervention. The proposed project, including the open trial and pilot RCT, will prepare us to conduct the next study in this line of research, i.e., a full-scale effectiveness study. Ultimately, we hope this will result in another tool to be used for suicide prevention in a high-risk clinical group.

#### F. Risk-Benefit Ratio

**Phase 1:** The risks to participants are judged to be acceptable relative to the anticipated benefits. Serious risks related to study participation are unlikely to occur. Benefits to the participant may include satisfaction with having a chance to tell one's story, talk about successful coping strategies, and potentially help other people.

Date most recently revised 3/22/2022

Protocol Version 2.5 

Phases 2 and 3: The risks to participants are judged to be acceptable relative to the anticipated benefits. Serious risks related to study participation are unlikely to occur. Benefits may include education if receiving the LifePlans intervention, and risk assessments and assistance obtaining appropriate treatment if needed at follow-up assessments.

# 4) REFERENCES

- 1. Houston TK, Cherrington A, Coley HL, et al. The art and science of patient storytelling-harnessing narrative communication for behavioral interventions: the ACCE project. *Journal of health communication*. Aug 2011:16(7):686-697.
- **2.** Houston TK, Allison JJ, Sussman M, et al. Culturally appropriate storytelling to improve blood pressure: a randomized trial. *Ann Intern Med.* Jan 18 2011;154(2):77-84.
- **3.** Gaudiano BA, Davis CH, Miller IW, Uebelacker LA. Development of a Storytelling Video Self-Help Intervention Based on Acceptance and Commitment Therapy for Major Depression: Open Trial Results. *Behav Modif.* Oct 1 2017:145445517738932.
- **4.** Gortner EM, Rude SS, Pennebaker JW. Benefits of expressive writing in lowering rumination and depressive symptoms. *Behavior therapy*. Sep 2006;37(3):292-303.
- **5.** Graf MC, Gaudiano BA, Geller PA. Written emotional disclosure: a controlled study of the benefits of expressive writing homework in outpatient psychotherapy. *Psychother Res.* Jul 2008;18(4):389-399.
- **6.** Devilly GJ, Borkovec TD. Psychometric properties of the credibility/ expectancy questionnaire. *Journal of Behavior Therapy and Experimental Psychiatry*. 2000;31:73-86.
- **7.** Larsen DL, Attkisson CC, Hargreaves WA, al. e. Assessment of client/ patient satisfaction: development of a general scale. *Evaluation and Program Planning*. 1979;2:197-207.
- **8.** Nguyen TD, Attkisson CC, Stegner BL. Assessment of patient satisfaction: development and refinement of a service evaluation questionnaire. *Evaluation and Program Planning*. 1983;6(299-313).
- **9.** Green MC, Brock TC. The role of transportation in the persuasiveness of public narratives. *Journal of Personality and Social Psychology*. Nov 2000;79(5):701-721.
- **10.** Ondersma SJ, Chase SK, Svikis DS, Schuster CR. Computer-based brief motivational intervention for perinatal drug use. *J Subst Abuse Treat*. Jun 2005;28(4):305-312.
- Posner K, Brown GK, Stanley B, et al. The Columbia-Suicide Severity Rating Scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults. *Am J Psychiatry*. Dec 2011;168(12):1266-1277.
- **12.** Posner K. C-SSRS Training. 2012.
- **13.** Miller IW, Norman WH, Bishop SB, Dow MG. The Modified Scale for Suicidal Ideation: reliability and validity. *J Consult Clin Psychol.* Oct 1986;54(5):724-725.
- **14.** Derogatis L. *The Brief Symptom Inventory (BSI): Administration, scoring and procedures manual.* Baltimore: Clinical Psychometric Research;1992.
- **15.** Sheehan DV. MINI: Mini International Neuropsychiatric Interview, English Version 7.0.2 for DSM-5. 2016.
- **16.** Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. *J Psychiatr Res.* Nov 1975;12(3):189-198.
- 17. World Health Organization. WHO DAS II. Disabiltiy Assessment Schedule. 2003; http://www.who.int/icidh/whodas/generalinfo.html. Accessed October 24, 2003.
- **18.** Novak SP, Colpe LJ, Barker PR, Gfroerer JC. Development of a brief mental health impairment scale using a nationally representative sample in the USA. *Int J Methods Psychiatr Res.* Jun 2010;19 Suppl 1:49-60.
- 19. Chwastiak LA, Von Korff M. Disability in depression and back pain. Evaluation of the World Health Organization Disability Assessment Schedule (WHO DAS II) in a primary care setting. *Journal of Clinical Epidemiology*. 2003;56:507-514.
- **20.** Batterham PJ, Calear AL, Christensen H. The Stigma of Suicide Scale. Psychometric properties and correlates of the stigma of suicide. *Crisis.* Jan 1 2013;34(1):13-21.
- **21.** Vaux A, Riedel S, Stewart D. Modes of Social Support: The Social Support Behaviors (SS-B) Scale. *American Journal of Community Psychology*. 1987;15:209-232.

- **22.** D'Zurilla T, Nezu A, Maydeu Olivares A. *Manual for the Social Problem Solving Inventory-revised.* North Tonawanda, NY: Multi-health Systems;1999.
- **23.** Wilson KG, Sandoz EK, Kitchens J, Roberts ME. The Valued Living Questionnaire: Defining and measuring valued action within a behavioral framework. *The Psychological Record*. 2010;60:249-272.
- **24.** Morisky DE, Green LW, Levine DM. Concurrent and predictive validity of a self-reported measure of medication adherence. *Med Care*. Jan 1986;24(1):67-74.
- 25. Linehan MM. *Therapist Interview*. University of Washington, Seattle, WA1987.
- **26.** Kraemer HC, Kupfer DJ. Size of treatment effects and their importance to clinical research and practice. *Biol Psychiatry*. Jun 1 2006;59(11):990-996.
- **27.** Kraemer HC, Mintz J, Noda A, Tinklenberg J, Yesavage JA. Caution regarding the use of pilot studies to guide power calculations for study proposals. *Arch Gen Psychiatry*. May 2006;63(5):484-489.
- **28.** Crabtree BF, Miller WL. Using codes and code manuals: a template organizing style of interpretation. In: Crabtree BF, Miller WL, eds. *Doing Qualitative Research, 2nd edition*. Thousand Oaks, CA: Sage Publications; 1999:163-177.
- **29.** Babor TF, Higgins-Biddle JC, Saunders JB, Monteiro MG. *AUDIT: The Alcohol Use Disorders Identification Test. Guidelines for use in primary care, 2nd edition.* World Health Organization;2001.
- **30.** Berman AH, Bergman H, Palmstierna T, Schlyter F. *DUDIT Manual: The Drug Use Disorders Identification Test, Version 1.0.* Stockholm: Karolinska Institutet, Department of Clinical Neuroscience; 2005.
- **31.** Bebbington P, Nayani T. The Psychosis Screening Questionnaire. *International Journal of Methods in Psychiatric Research.* 1995;5:11-19.

| 5) CRITERIA FOR WAIVER OF AUTHORIZATION FOR USE OF PROTECTED HEALTH INFORMATION (PHI) |
|---|
| 5A. Does the requested use of PHI involve more than minimal risk to privacy? State of PHI involve more than minimal risk to privacy? State of PHI waiver] NO [if "NO," address 1-3 below] |
| 1. Plan to Protect Patient Identifiers from Improper Use and Disclosure: Potential risks due to loss of confidentiality will be minimized by having all information collected and handled by research staff trained to deal appropriately with sensitive clinical issues. All research personnel will receive training in research ethics and be approved by the institution to conduct research. All information will be kept in locked files. Electronic data will be stored on encrypted drives/servers and password protected. Data will be available only to authorized personnel and subject codes will be used to store information in databases. No subject will be identified in any report of this project. |
| <ol> <li>Plan to Destroy Identifiers or Justification for Retaining Identifiers:</li> <li>PHI will be destroyed upon study completion plus 1 year.</li> </ol> |
| 3. Assurances that the PHI will not be Re-used or Disclosed: Information collected will only be used for the purposes described below and will be treated as confidential material as described above. |
| 5B. Could the research be practicably conducted without a waiver? ☐ YES ☐ NO 5C. Could the research be practicably conducted without access to and use of the PHI? ☐ YES ☐ NO 5D. PHI is only needed for activities preparatory to research ☐ YES ☐ NO |
| 6) DESCRIPTION OF PHI TO BE COLLECTED UNDER WAIVER |

Chart reviews of new patients will be routinely conducted by study staff to determine if they are likely to meet inclusion/exclusions criteria for the study as described above. PHI to be obtained: patient demographic and contact information (name, address, telephone numbers, gender, age, race, marital status, occupation status) and patient psychiatric/treatment history (diagnoses and suicide history, past and current psychological and/or pharmacological treatments, current mental health provider contact information, lab results).

Date most recently revised 3/22/2022

Protocol Version 2.5 

# 7) ADVERTISEMENTS

Document attached.

# 8) INFORMED CONSENT FORM (ICF), ASSENT OF MINOR & PARENTAL PERMISSION FORM

# Indicate number of consent(s): 9

# Identify each consent (i.e., Main, Screening, DNA):

- Verbal Consent for email and videorecording prior to enrollment
- Phase 1A Written consent
- Phase 1A-- Verbal consent
- Phase 1B- Consent for use of videos in LifePlans intervention
- Phase 1B HIPAA release; media release; materials release; COVID risk acknowledgment
- Phase 2 Main Written consent
- Phase 2 Stakeholders Written consent
- Phase 3 Written consent
- Phase 3 Email/Videoconferencing verbal consent